CLINICAL TRIAL: NCT01490073
Title: The Effect of Nitroglycerin on the IUD Insertion Experience in Nulliparous Women: a Pilot Study
Brief Title: The Effect of Nitroglycerin on the Intrauterine Device (IUD) Insertion Experience in Nulliparous Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: American College of Obstetricians and Gynecologists (Other); Bayer (Industry)
Responsible Party: Principal Investigator, Elizabeth Micks, Instructor and Fellow in Family Planning, Department of Obstetrics and Gynecology, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 7928
Record Dates: First submitted 2011-12-08; First posted 2011-12-12 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Contraception; Pain
Keywords: Intrauterine device; Pain; Contraception; Nitroglycerin; Nitric oxide donor; Intrauterine device insertion
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active nitroglycerin ointment (Active Comparator)
  Interventions: Drug: Insertion of nitroglycerin ointment
- Placebo ointment (Placebo Comparator)
  Interventions: Drug: Insertion of placebo ointment

INTERVENTIONS:
Drug: Insertion of nitroglycerin ointment — Nitroglycerin ointment inserted into the vagina 30-45 minutes prior to IUD insertion
  Arms: Active nitroglycerin ointment
Drug: Insertion of placebo ointment — Placebo ointment inserted into the vagina 30-45 minutes prior to IUD insertion
  Arms: Placebo ointment

SUMMARY:
Increasing ease of access of long-acting birth control methods, like intrauterine devices (IUDs), is an important way to reduce the risk of unintended pregnancy. Unfortunately, fear of IUD insertion in women who have not had children is common among health care providers and women alike, and this limits IUD use. To increase acceptance of this highly effective birth control method, there is a need to explore new, low cost, and easily applied methods to improve the insertion experience. This is a pilot study to evaluate the effectiveness and acceptability of nitroglycerin ointment applied vaginally to improve the IUD insertion experience for both patient and provider. The investigators hypothesis is that nitroglycerin ointment will decrease the pain associated with IUD insertion.

DETAILED DESCRIPTION:
Increasing acceptability and use of long acting reversible contraceptive methods like the intrauterine device (IUD) is an important strategy to reduce the risk of unintended pregnancy. Unfortunately, fear of IUD insertion in nulliparous women is common among health care providers and women alike, and this limits IUD use. While many health care providers assume that placement is more difficult in nulliparous women, there is no evidence that the risk of unsuccessful insertion is higher. Women worry about pain with insertion, and their fear is not unfounded as U.S. and international data have shown that nulliparous women report approximately twice as much pain with IUD insertion compared to parous women.

A key difference between nulliparous and multiparous women is the resistance of the cervix. While cervical dilation is uncommonly needed during IUD placement, force is often required to pass the insertion device through the internal os. Although misoprostol and ibuprofen have been studied as ways to improve the IUD insertion experience, neither has proved effective, and misoprostol actually has been shown to increase pain. Therefore, to increase acceptance of this highly effective contraceptive, there is a need to investigate novel, low cost, easily applied and accessible techniques to improve the insertion experience.

Nitric oxide (NO) donors, including nitroglycerin, nitroprusside, isosorbide mononitrate and isosorbide dinitrate, have effects on the animal and human cervix. Both nitroglycerin and isosorbide mononitrate tablets administered vaginally have been shown in RCTs to induce effective cervical ripening with minimal side effects for first trimester abortion compared to placebo. Nitroprusside and isosorbide dinitrate gel given intracervically prior to first trimester abortion also have showed minimal side effects in several RCTs, but with mixed results regarding effectiveness. Additional safety data about NO donors applied topically to skin and mucosal surfaces is well established through the routine use of topical nitroglycerin for treatment of anal fissures.

Although a recent randomized controlled trial (RCT) comparing nitroprusside gel to misoprostol for cervical ripening prior to first trimester surgical abortion found superior cervical dilation in the misoprostol group, there was no significant difference in cervical dilation up to 5 mm. While most studies of abortion are concerned with providing adequate dilation beyond 8 mm, the cervical remodeling that is necessary to help with IUD insertion is much less, as the levonorgestrel intrauterine system (LNG-IUS) inserter is only 4.75 mm in diameter. Since NO donors are smooth muscle relaxants, they are expected to induce cervical ripening without causing uterine cramping, which is the most significant side effect of misoprostol.

Nitroglycerin is inexpensive, stable at room temperature, and readily available in tablet and ointment form, as well as in a dextrose solution for intravenous administration. The ointment form is commonly applied topically for the treatment of anal fissures. We propose the following aims:

1. To determine if nitroglycerin ointment applied vaginally 30-45 minutes prior to IUD insertion improves pain among nulliparous women compared to a placebo ointment. Self-reported pain scores on a 100 mm VAS will be assessed at multiple time points during and after the IUD insertion procedure. In addition, overall satisfaction and adverse effects will be evaluated.
2. To determine if nitroglycerin ointment applied vaginally 30-45 minutes prior to IUD insertion improves ease of IUD insertion for the provider compared to a placebo ointment. In addition, need for additional dilation, additional pain medicine such as paracervical block, inability to place the IUD, and complications will be tracked.
3. To determine if nitroglycerin ointment applied vaginally 30-45 minutes prior to IUD insertion is safe and well tolerated. Side effects related to treatment with nitroglycerin ointment or placebo will be compared. Blood pressure will be measured at multiple time points.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-45 years,
2. generally healthy,
3. requesting a LNG-IUS for contraception as the primary indication

Exclusion Criteria:

1. Previous pregnancy beyond 20 weeks;
2. previous IUD placement or attempted IUD placement;
3. previous cervical cold knife cone (CKC) or loop electrosurgical excision procedure (LEEP);
4. contraindication to LNG-IUS (including pregnancy, fibroids that distort the uterine cavity, exam consistent with PID, allergy to any component of the LNG-IUS, etc);
5. concurrent use of any form of nitrate therapy or medications that interact with nitroglycerin (such as phosphodiesterase V inhibitors);
6. known allergy to nitroglycerine or common topical ointment ingredients;
7. known renal or hepatic impairment;
8. history of hypertensive or hypotensive disorder;
9. history of migraine, cluster headaches, or vascular headaches;
10. history of myocardial infarction;
11. uncontrolled congestive heart failure;
12. unstable angina;
13. tobacco or alcohol amblyopia;
14. congenital optic atrophy;
15. blood pressure less than 90/55 or greater than 150/100 in office prior to speculum exam

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2012-11-01 (Actual); Study Completion 2012-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Planned Parenthood Columbia Willamette, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Nitroglycerin Ointment | Placebo Ointment
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Nitroglycerin Ointment | Placebo Ointment | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (6.9) | 25.7 (4.4) | 27.04 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 9 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Current smoker [Count of Participants; unit: Participants] | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Patient-reported Pain at Passage of Insertion Device Through Cervix, as Measured on a 100 mm VAS
Description: Patient-reported pain at passage of insertion device through cervix, as measured on a 100 mm VAS. VAS anchors: 0 indicates no pain, and 100 indicates worst pain imaginable.
Time Frame: 30-45 minutes after insertion of nitroglycerin ointment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Active Nitroglycerin Ointment | Placebo Ointment
Number analyzed (Participants) | 12 | 12
mm | 55.8 (25.2) | 53.9 (28.1)

2. Secondary Outcome: Provider Ease With Intrauterine Device Insertion Measured on a 100 mm VAS
Description: Provider ease with intrauterine device insertion measured on a 100 mm VAS. VAS (visual analog scale) anchors: 0 indicates easiest insertion imaginable, 100 indicates most difficult insertion imaginable
Time Frame: 30-45 minutes after insertion of nitroglycerin ointment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Active Nitroglycerin Ointment | Placebo Ointment
Number analyzed (Participants) | 12 | 12
mm | 29.4 (23.8) | 22.8 (29.9)

ADVERSE EVENTS:
Time Frame: 2 days
Description: Subjects were asked about the presence of side effects including headache, lightheadedness, palpitations, nausea, vomiting, cramping and diarrhea. Discomfort or irritation from the vaginal ointment was also assessed. Subjects were contacted approximately 24 h after IUD insertion and asked about side effects or other new medical concerns or events during the postprocedure interval.
Arm/Group | Active Nitroglycerin Ointment | Placebo Ointment
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No